CLINICAL TRIAL: NCT07202000
Title: Double-blind, Prospective, Randomized, Placebo-controlled Trial to Assess if Activin Ligand-trap Biological Therapy Can Improve Exercise Capacity and Cognitive Function in Heart Failure With Preserved Ejection Fraction Compared to Placebo.
Brief Title: EXercise and Activin Inhibition to Modulate InflammatioN Effects on Heart Failure and Cognition (EXAMINE-HFC)
Acronym: EXAMINE-HFC
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: American Heart Association (Other); University of Michigan (Other); Oakland University (Other)
Responsible Party: Principal Investigator, Gregory D. Lewis, M.D., Professor of Medicine, Massachusetts General Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2024P001990
Record Dates: First submitted 2025-09-08; First posted 2025-10-01 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Heart Failure With Preserved Ejection Fraction
Keywords: heart failure with preserved ejection fraction; exercise capacity; activin inhibition; cognition
MeSH Terms: interventions — Saline Solution

STUDY DESIGN:
Intervention Model Description: Double-blind, prospective, phase 2 randomized, placebo-controlled 24-week clinical trial with a crossover at week 12.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Activin ligand-trap biological therapy (KER-012) subcutaneously (SC) 1.5mg/kg every 4 weeks X 3 (Active Comparator): Activin ligand-trap biological therapy subcutaneously in addition to an individualized physical activity program for 12 weeks before the crossover.
  Interventions: Drug: Activin ligand-trap biological therapy
- Normal Saline subcutaneous injection every 4 weeks X 3 (Placebo Comparator): Patients will receive placebo in addition to an individualized physical activity program for 12 weeks before the crossover.
  Interventions: Drug: Placebo, Normal Saline

INTERVENTIONS:
Drug: Activin ligand-trap biological therapy — Investigational therapy
  Arms: Activin ligand-trap biological therapy (KER-012) subcutaneously (SC) 1.5mg/kg every 4 weeks X 3
Drug: Placebo, Normal Saline — Inactive drug
  Arms: Normal Saline subcutaneous injection every 4 weeks X 3

SUMMARY:
The goal of this clinical trial is to learn if therapy with activin ligand-trap biological therapy (an investigational drug) combined with exercise training can improve exercise capacity and cognitive function in heart failure with preserved ejection fraction (HFpEF). The main questions it aims to answer are:

* Does activin-ligand trap biological therapy improve exercise capacity as measured by change in peak oxygen uptake (peak VO2) from baseline to week 12?
* Does activin-ligand trap biological therapy improve cognitive function as assessed by the NIH-Toolbox Cognition Battery (NIHTB-CB) composite score and Rey Auditory Verbal Learning Test (RAVLT) from baseline to week 12?

Researchers will compare activin-ligand trap biological therapy to a placebo (a look-alike substance that contains no drug) to see if activin-ligand trap therapy works to improve exercise capacity and cognitive function in patients with HFpEF.

DETAILED DESCRIPTION:
A double-blind, prospective, phase 2 randomized, placebo-controlled 24-week clinical trial to assess exercise tolerance after activin-ligand trap biological therapy compared to placebo in HFpEF patients with a primary endpoint of change in peak VO2.

Forty-eight participants with HFpEF who are overweight or obese will be recruited from the Cardiopulmonary Exercise Testing (CPET) Laboratory and will have a recent or scheduled clinical care CPET. These measurements will serve as baseline measures. After undergoing other baseline measurements such as actigraphy, blood studies, DEXA scan, Kansas City Cardiomyopathy Questionnaire (KCCQ), NIHTB-CB, and RAVLT, participants will be randomized (1:1) to either activin-ligand trap biological therapy combined with physical activity (n=24) or placebo combined with physical activity (n=24). Randomization will be stratified by sex and will be performed in permutated blocks of 4 to assure balanced group sizes. In order to allocate without bias and in a manner blinded to both participants and investigators, we will use random number generation at the time of randomization. After 12 weeks, patients will return for a new CPET, physical exam, urine and blood test, echocardiogram, electrocardiogram, DEXA scan, actigraphy, assessment of NYHA class, NIHTB-CB, RAVLT, KCCQ, six-minute walk test, handgrip test, and adverse events assessment. After these assessments, patients will undergo crossover at week 12 and will receive either the activin-ligand trap biological therapy combined with physical activity (n=24) or the placebo combined with physical activity (n=24) for an additional 12 weeks. At week 24, patients will return to have a repeat of the same tests that were performed at week 12.

ELIGIBILITY:
Inclusion Criteria:

1. Adult ≥ 40 years of age;
2. Body mass index ≥ 27 kg/m2;
3. Left ventricular ejection fraction (LVEF) ≥ 0.50 with NYHA II-III;
4. Established diagnosis of HFpEF based on medical history supported by at least one of the following 5 criteria (i through v, below)

   i. Documented hospitalization with HFpEF as a primary cause or other urgent outpatient visit for acute HFpEF (as primary cause) at which IV loop diuretic was provided as treatment (≥ 1 month prior to screening);

   ii. Increased left atrial (LA) size: AP dimension: ≥ 4.0 in men, > 3.8 in women; or LA length ≥ 5.0 cm or LA volume ≥ 55 mL or LA volume index≥ 29 mL/m2;

   iii. PCWP at rest > 15 mmHg (or LVEDP ≥ 18 mmHg) or ≥ 25 mmHg with exercise (or PCWP/CO ≥ 2.0 mmHg/L/min with exercise);

   iv. Either of the following at rest by Doppler and Tissue Dopper: a) for patients in sinus rhythm: E/e' ratio ≥ 15 at septal annulus, or E/e' ratio ≥ 13 at lateral annulus, or average E/e' ratio ≥ 14; for patients in atrial fibrillation E/e' ≥ 11 at the septal annulus;

   v. Elevated NT-proBNP ≥ 125 pg/mL (≥ 250 with chronic atrial fibrillation).
5. Achievement of a respiratory exchange ratio (RER) at baseline CPET of ≥ 1.05 to ensure maximum volitional effort was provided;
6. Ambulatory (not wheelchair/scooter-dependent) and able to perform CPET/6MWT/Chair stand evaluations;
7. Stable dose of medications (defined as no new medication or change in existing dose of medication ≥ 50%) for at least 30 days prior to screening.

Exclusion Criteria:

1. Conditions anticipated to independently impact exercise capacity or clinical stability during the trial period

   1. Current or recent (within 30 days) acute decompensated HF requiring intravenous diuretics or hospitalization;
   2. Initiation of treatment with GLP-1 receptor agonist or SGLT2 inhibitor within 60 days of screening;
   3. Planned cardiac surgery or catheter intervention during the period of trial participation;
   4. Entry within 30 days of screening or plans to enter a weight loss program and/or cardiac rehabilitation or initiate any new exercise program during the study.
2. Primary cardiomyopathy (e.g., constrictive, restrictive, infiltrative, toxic, hypertrophic, congenital), LVEF < 40% within the last 3 years, or active myocarditis;
3. Lactating, pregnant, or planning to become pregnant;
4. Non-cardiac organ system dysfunction or sufficient severity to predominate as the source of exercise intolerance in addition to the following specific criteria: pulmonary disease with chronic home daytime supplemental O2 dependence, severe anemia with hemoglobin < 9 g/dL or chronic kidney disease (CKD) with estimated GFR < 30 mL/min/1.73m2 based on the CKD-EPI equation.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2027-07 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Change in peak oxygen uptake (peak VO2) in HFpEF subjects following activin ligand-trap biological therapy or placebo. | From baseline to week 12 and from week 12 to week 24
  Peak VO2 measured by a maximal effort Cardiopulmonary Exercise Test (CPET).

SECONDARY OUTCOMES:
Change in cognitive function. | From baseline to week 12 and from week 12 to week 24
  Changes in cognitive function as assessed by the NIH-Toolbox Cognition Battery (NIHTB-CB) composite score standardized by age.
Change in cognitive function | From Baseline to week 12, and from week 12- 24
  changes in cognitive function as assessed by comparing the Rey Auditory Verbal Learning Test (RAVLT) score, standardized by age.
Change in body composition. | From baseline to week 12 and week 12 to week 24
  Change in body composition as measured by DEXA scan to compare the % lean muscle mass and absolute quantity of lean muscle mass
Change in cardiac function measured by echocardiography | From baseline to week 12 and from week 12 to 24
  Change in Left Atrium (LA)dimensions (cm)
Change in cardiac function measured by echocardiography | From baseline to week 12 and from week 12 to week 24
  Change in E/e' ratio
Change in patient-reported Quality of Life . | From baseline to week 12 and from week 12 to 24
  Change to Quality of Life as measured by the Kansas City Cardiomyopathy Questionnaire score
Change in New York Heart Association (NYHA) Functional Class. | From baseline to week 12 and week 12 - 24
  Change in New York Heart Association (NYHA) classification system which categorizes heart failure severity into four classes based on physical activity limitations and symptoms.
  Class I :No limitation of physical activity; Class II: Slight limitation of physical activity; Class III:Marked limitation of physical activity; Class IV: Unable to carry on any physical activity without discomfort; symptoms of heart failure at rest
Change metabolic measures such as in Hemoglobin A1C (HbA1C) | From baseline to week 12, and week 12 to week 24
  Change in HbA1C
Changes in metabolic measures such as waist to hip measurements | From baseline to week 12 and week 12 to week 24
  Change in waist-to-hip ratio
Change in six-minute walk distance | From baseline to week 12 and week 12 -24
  percent change in six-minute walk distance (6MWD)
Change in physical activity as measured by the Apple Health App | From baseline to week 12 and week 12 to weeks 24
  Percent change in physical activity as measured by the Apple Health App
Changes in cardiovascular risk biomarkers: high sensitivity c-Reactive Protein (hs-CRP) | From baseline to week 12 and from week 12 to week 24
  Change in high sensitivity c-Reactive Protein (hs-CRP) (ml/L)
Change in cardiovascular biomarkers: N-terminal pro-B-type natriuretic peptide (NTproBNP) | from baseline to week 12 and from week 12 week 24
  Change in N-terminal pro-B-type natriuretic peptide (NTproBNP) (pg/ml)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory D. Lewis, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nayor M, Houstis NE, Namasivayam M, Rouvina J, Hardin C, Shah RV, Ho JE, Malhotra R, Lewis GD. Impaired Exercise Tolerance in Heart Failure With Preserved Ejection Fraction: Quantification of Multiorgan System Reserve Capacity. JACC Heart Fail. 2020 Aug;8(8):605-617. doi: 10.1016/j.jchf.2020.03.008. Epub 2020 Jun 10. PMID 32535122
- [Background] Roh JD, Hobson R, Chaudhari V, Quintero P, Yeri A, Benson M, Xiao C, Zlotoff D, Bezzerides V, Houstis N, Platt C, Damilano F, Lindman BR, Elmariah S, Biersmith M, Lee SJ, Seidman CE, Seidman JG, Gerszten RE, Lach-Trifilieff E, Glass DJ, Rosenzweig A. Activin type II receptor signaling in cardiac aging and heart failure. Sci Transl Med. 2019 Mar 6;11(482):eaau8680. doi: 10.1126/scitranslmed.aau8680. PMID 30842316
- [Background] Houstis NE, Eisman AS, Pappagianopoulos PP, Wooster L, Bailey CS, Wagner PD, Lewis GD. Exercise Intolerance in Heart Failure With Preserved Ejection Fraction: Diagnosing and Ranking Its Causes Using Personalized O2 Pathway Analysis. Circulation. 2018 Jan 9;137(2):148-161. doi: 10.1161/CIRCULATIONAHA.117.029058. Epub 2017 Oct 9. PMID 28993402
- [Background] Dhakal BP, Malhotra R, Murphy RM, Pappagianopoulos PP, Baggish AL, Weiner RB, Houstis NE, Eisman AS, Hough SS, Lewis GD. Mechanisms of exercise intolerance in heart failure with preserved ejection fraction: the role of abnormal peripheral oxygen extraction. Circ Heart Fail. 2015 Mar;8(2):286-94. doi: 10.1161/CIRCHEARTFAILURE.114.001825. Epub 2014 Oct 24. PMID 25344549
- [Background] Callaghan BC, Reynolds EL, Banerjee M, Chant E, Villegas-Umana E, Gardner TW, Votruba K, Giordani B, Pop-Busui R, Pennathur S, Feldman EL. The Prevalence and Determinants of Cognitive Deficits and Traditional Diabetic Complications in the Severely Obese. Diabetes Care. 2020 Mar;43(3):683-690. doi: 10.2337/dc19-1642. Epub 2020 Jan 13. PMID 31932459
- [Background] Hammond CA, Blades NJ, Chaudhry SI, Dodson JA, Longstreth WT Jr, Heckbert SR, Psaty BM, Arnold AM, Dublin S, Sitlani CM, Gardin JM, Thielke SM, Nanna MG, Gottesman RF, Newman AB, Thacker EL. Long-Term Cognitive Decline After Newly Diagnosed Heart Failure: Longitudinal Analysis in the CHS (Cardiovascular Health Study). Circ Heart Fail. 2018 Mar;11(3):e004476. doi: 10.1161/CIRCHEARTFAILURE.117.004476. PMID 29523517
- [Background] Ho JE, Zern EK, Wooster L, Bailey CS, Cunningham T, Eisman AS, Hardin KM, Zampierollo GA, Jarolim P, Pappagianopoulos PP, Malhotra R, Nayor M, Lewis GD. Differential Clinical Profiles, Exercise Responses, and Outcomes Associated With Existing HFpEF Definitions. Circulation. 2019 Jul 30;140(5):353-365. doi: 10.1161/CIRCULATIONAHA.118.039136. Epub 2019 May 28. PMID 31132875